CLINICAL TRIAL: NCT04468035
Title: Early Cognitive Assessment and Evolutionary Monitoring of Patients With Severe ARDS (Acute Respiratory Distress Syndrome) on SARS-CoV2 Viral Pneumonia Requiring Mechanical Ventilation
Brief Title: Early Cognitive Assessment and Evolutionary Monitoring of Patients With Severe ARDS on COVID-19 Pneumonia Requiring Mechanical Ventilation
Acronym: CognitiVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CognitiVID
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The new coronavirus pandemic responsible for the severe acute respiratory syndrome SARS-CoV2 requires, in its severe forms, the use of invasive ventilation in intensive care.

The first patients seen in intensive care presented with neurological symptoms and usually not seen in non-viral ARDS or due to other viral causes. These were mainly restless awakenings, attempts at self-extubation and confusional syndromes. Although the data in the literature do not seem to reveal the presence of SARS-CoV2 in the CSF of these patients, certain elements seem to show parenchymal brain damage with the description of hypometabolism of the frontal regions. In addition, most of these patients present a memory complaint after going into intensive care (personal data not published).

We do not know to date what is the cognitive and psychic profile of these patients, nor what will be their future evolution. Some patients may require specific neuro-cognitive rehabilitation.

The aim of this study is to assess the cognitive profile of patients infected with COVID-19 who have used invasive ventilation in the intensive care unit of Paris Saint-Joseph hospital since April 2020, in order to be able to compare them between them and follow their evolution in the medium term. This work could make it possible to describe the specific cognitive impairment of SARS-CoV2, by trying to evade other causes of cognitive disorders in patients hospitalized in intensive care for respiratory distress (hypoxia, treatments, metabolic disorders, etc.).

The main objective is to follow the medium-term evolution between 3 and 6 months of the cognitive profile of patients with severe form of SARS-CoV2 with the use of ventilatory resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with SARS-CoV2 treated in the intensive care unit of the HPSJ for respiratory distress, using invasive ventilation by oro-tracheal intubation from April 2020
* French speaking patient

Exclusion Criteria:

* Patient with an alertness disorder with Glasgow eye score <3 and / or motor <6 (confusion being a poor criterion for evaluating the Glasgow score apart from head trauma).
* Patient with impossibility to communicate (mutism, aphonia, major language barrier)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit of the Paris Saint-Joseph Hospital (HPSJ), for the management of their respiratory distress following COVID infection, between April 2020 and April 2021.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Medium-term evolution between 3 and 6 months | Month 6
  This ouctome corresponds to the medium-term evolution between 3 and 6 months of the cognitive profile of patients with severe form of SARS-CoV2 with recourse to ventilatory resuscitation.

SECONDARY OUTCOMES:
Cognitive impairment at M3 | Month 3
  This outcome corresponds to MMSE orientation score.
Cognitive impairment at M6 | Month 6
  This outcome corresponds to MMSE orientation score.
Memory Scores at M3 | Month 3
  This outcome corresponds to Memory scores.
Memory Scores at M6 | Month 6
  This outcome corresponds to Memory scores.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Vialatte de Pémille, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Alkeridy WA, Almaghlouth I, Alrashed R, Alayed K, Binkhamis K, Alsharidi A, Liu-Ambrose T. A Unique Presentation of Delirium in a Patient with Otherwise Asymptomatic COVID-19. J Am Geriatr Soc. 2020 Jul;68(7):1382-1384. doi: 10.1111/jgs.16536. Epub 2020 May 16. PMID 32383778
- [Background] Helms J, Kremer S, Merdji H, Clere-Jehl R, Schenck M, Kummerlen C, Collange O, Boulay C, Fafi-Kremer S, Ohana M, Anheim M, Meziani F. Neurologic Features in Severe SARS-CoV-2 Infection. N Engl J Med. 2020 Jun 4;382(23):2268-2270. doi: 10.1056/NEJMc2008597. Epub 2020 Apr 15. No abstract available. PMID 32294339
- [Background] Bouattour N, Farhat N, Hadjkacem H, Hdiji O, Sakka S, Dammak M, Mhiri C. [Five-word test calibration in a Tunisian population of healthy subjects]. Pan Afr Med J. 2019 Sep 30;34:58. doi: 10.11604/pamj.2019.34.58.14472. eCollection 2019. French. PMID 31762923
- [Background] Maillet D, Matharan F, Le Clesiau H, Bailon O, Peres K, Amieva H, Belin C. TNI-93: A New Memory Test for Dementia Detection in Illiterate and Low-Educated Patients. Arch Clin Neuropsychol. 2016 Dec 1;31(8):896-903. doi: 10.1093/arclin/acw065. PMID 27590305
- [Result] Vialatte de Pemille C, Ray A, Michel A, Stefano F, Yim T, Bruel C, Zuber M. Prevalence and prospective evaluation of cognitive dysfunctions after SARS due to SARS-CoV-2 virus. The COgnitiVID study. Rev Neurol (Paris). 2022 Oct;178(8):802-807. doi: 10.1016/j.neurol.2022.03.014. Epub 2022 May 13. PMID 35610098